CLINICAL TRIAL: NCT01448005
Title: Post-market Release Registry of Wearable Defibrillator Use in Patients With Ventricular Dysfunction Following CABG Surgery
Brief Title: LifeVest Post-CABG Registry
Status: Terminated | Type: Observational
Why Stopped: Enrollment
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0107
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Sudden Cardiac Death; Ventricular Fibrillation; Ventricular Tachycardia; Ventricular Dysfunction; Myocardial Ischemia
Keywords: Coronary Artery Bypass Grafting; Resuscitation; Sudden Cardiac Death; Ventricular Dysfunction
MeSH Terms: conditions — Death, Sudden, Cardiac; Ventricular Fibrillation; Tachycardia, Ventricular; Ventricular Dysfunction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- wearable defibrillator use: subjects will use a wearable defibrillator
  Interventions: Device: wearable defibrillator (LifeVest)

INTERVENTIONS:
Device: wearable defibrillator (LifeVest) — A wearable defibrillator automatically detects and treats ventricular tachycardia and ventricular fibrillation without the need for bystander intervention.
  Other Names: LifeVest; wearable cardioverter defibrillator; wearable automatic external defibrillator

SUMMARY:
This is a multi-center prospective registry of patients with an ejection fraction (EF) ≤ 35% following coronary artery bypass graft (CABG) surgery in order to test the hypothesis that wearable defibrillators (WD) will decrease overall mortality after discharge by decreasing arrhythmic death in this select population with high risk for sudden cardiac death (SCD). This is a pilot project to determine the feasibility of a larger-scale study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone CABG surgery during current hospitalization
* Patients who have an ejection fraction ≤ 35% following the surgery.
* Patients who have dilated cardiomyopathy or prior myocardial infarction.
* Patients who are prescribed a wearable defibrillator following surgery.
* Patient who are at least 18 years old.

Exclusion Criteria:

* Patients who have an active ICD.
* Patients who have an active unipolar pacemaker.
* Patients having a chest circumference over 56 inches or under 26 inches.
* Patients who are unable to consent or unwilling to wear the WCD after discharge or who do not agree to be contacted at 90 days.
* Patients with a mental, visual, physical or auditory deficit that could impair their ability to properly interact with a wearable defibrillator.
* Patients participating in another clinical study with mortality as the primary endpoint.
* Patients unable to use a wearable defibrillator due to physical conditions (bandages preventing electrode contact, physical deformities preventing electrode contact, dextrocardia, etc.).
* Patients who have decided to forgo resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone CABG surgery during current hospitalization and have an ejection fraction ≤ 35% following the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
number of patients who experience sudden cardiac death | three months

SECONDARY OUTCOMES:
number of patients who experience inappropriate shocks | three months
hours per day of wearable defibrillator use | three months
number of patients who experience sudden cardiac arrest | three months

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Szymkiewicz, MD, Study Director — Zoll Medical Corporation
Locations (5):
- United States (5):
  - Sutter Heart and Vascular Institute, Sacramento, California
  - Saint Joseph's Health System, Inc., Atlanta, Georgia
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Texas Heart Institute, St. Luke's Episcopal Hospital, Houston, Texas
  - Chippenham Johnston-Willis Medical Center, Richmond, Virginia